CLINICAL TRIAL: NCT04578132
Title: Observational Retrospective-prospective Study in Patients With Genitourinary Tumors Presenting COVID-19 Infection (SOGUG-COVID-19)
Brief Title: Description of the Population With Genitourinary Tumors and COVID-19
Acronym: SOGUGCOVID
Status: Completed | Type: Observational
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Responsible Party: Sponsor
Other Study IDs: SOG-INM-2020-04
Record Dates: First submitted 2020-10-06; First posted 2020-10-08 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Genito Urinary Cancer
Keywords: Urothelial cancer; prostate cancer; Germ line cancer; Kidney cancer; COVID-19
MeSH Terms: conditions — COVID-19; Urogenital Neoplasms; Prostatic Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genitourinary cancer patients that suffered COVID-19: Patients diagnosed with genitourinary cancer (urothelial, kidney, prostate and germ) that suffered from COVID-19 infection prior to cancer treatment, during treatment, or after treatment.

SUMMARY:
The identification of patients with genitourinary tumors who suffer from the infection by the Serious Acute Respiratory Syndrome Corona-Virus 2 (SARS-CoV-2) virus can represent multiple benefits both for themselves and for health professionals and the health system itself. We would be able to know more precisely the clinical evolution of these type of patient, to know their prognosis and being capable to select the most appropriate treatment modality for future pandemics.

SOGUG-COVID is an observational prospective-retrospective trial purely epidemiological, that aims to describe the population with genitourinary tumors (urothelial cancer, prostate cancer, testicular cancer and kidney cancer) infected by COrona VIrus Disease 19 (COVID-19) treated in Spanish hospitals, learn about the clinical presentation, therapeutic evolution and prognosis of said intercurrent infectious process, as well as its possible relationship with different clinical and therapeutic factors.

DETAILED DESCRIPTION:
The study will be carried out in Spanish hospitals, with principal investigators belonging to the medical oncology services of the SOGUG group (Spanish Group of Genitourinary Oncology), who will act as promoter. Once the patients have been selected, the variables of interest will be collected and studied. The main variables to record will be:

1. Patient characteristics
2. Hospital center where the patient is recruited
3. Pathological history:

   Concomitant pathology Usual drug treatment
4. Tumor pathology:

   Tumor type, histology, and stage (initial and at diagnosis of infection) Cancer diagnosis date Active cancer treatment or follow-up Participation in clinical trial Type of treatment most recently received for the infection (Surgery; Radiotherapy; Chemotherapy, Immunotherapy ...) Treatment lines, initiation and last dose received of the most recent most recent cancer treatment
5. COVID-19 infection:

   Confirmation date of COVID-19 infection PCR (Polymerase Chain Reaction) diagnostic test Immunoglobulin G (IgG) or Immunoglobulin M (IgM) serological diagnostic test Present symptoms, analytical alterations, thrombosis associated with COVID-19 infection, complications of infection Date of onset and disappearance of symptoms Days of fever and cough Radiological examination at the time of greatest severity Treatments received for COVID-19 Status upon discharge Date of discharge / exitus Negative presence of virus by PCR and PCR date
6. For patients who are receiving or have received immunotherapy treatments, additional information will be collected:

   Immunotherapy treatment line and type Start / end date and last dose previous infection of the treatment with immunotherapy Adverse effects
7. Prospective follow-up data (6 months from patient inclusion):

Date of start or restart of cancer treatment after infection Change / suspension of cancer treatment after COVID-19 Date of surgery in neoadjuvant patients Recurrence of COVID-19 Best response obtained Date of progression to cancer treatment Current status and date of last contact The study will use the data obtained from the patient's medical history, with no plans to use other sources.

The assignment of a patient to a specific therapeutic strategy has already been decided in advance by the usual clinical practice of medicine; The decision to prescribe a specific treatment is clearly dissociated from the decision to include a patient in the study. No intervention will be applied to patients, whether diagnostic or follow-up, that is not the usual clinical practice. Epidemiological methods will be used to analyze the collected data.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old.
* Diagnosed with genitourinary cancer (urothelial, kidney, prostate and germ).
* COVID-19 infection prior to cancer treatment, during treatment, or after treatment.
* The COVID-19 infection must be confirmed by PCR or serology, regardless of whether or not the patient requires hospitalization for the infection, additionally, a clinical and / or radiological determination must be available in those patients who present symptoms.

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with genitourinary cancer (urothelial, kidney, prostate and germ) that suffered COVID-19 infection prior to cancer treatment, during treatment, or after treatment.
Sampling Method: Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Ángel Climent, M.D., Ph.D., Study Chair — Instituto Valenciano de Oncología; Javier Puente, M.D., Ph.D., Study Chair — Hospital Clínico San Carlos de Madrid; Aránzazu González del Alba, M.D., Ph.D., Study Chair — Hospital Universitario Puerta de Hierro-Majadahonda; Sergio Vázquez Estevez, M.D., Ph.D., Study Chair — Hospital Universitario Lucus Augusti; Natalia Vidal, M.D., Ph.D., Study Chair — Hospital Clínico San Carlos de Madrid
Locations (32):
- Spain (32):
  - Institut Català d'Oncologia L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Althaia, Manresa, Barcelona
  - Hospital Universitari Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda, Madrid
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital del Mar, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d Hebron, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofía, Córdoba
  - Instituto Catalán de Oncología- Girona, Girona
  - Hospital Universitario Lucus Augusti, Lugo
  - Fundación Jiménez Díaz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico San Carlos de Madrid, Madrid
  - Hospital Infanta Leonor,, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Quironsalud, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Complejo Hospitalario Universitario Ourense, Ourense
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Nuestra Señora del Prado, Talavera de la Reina
  - Hospital Virgen de la Salud, Toledo
  - Hospital Universitario Dr. Peset, Valencia
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Txagorritxu, Vitoria-Gasteiz
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Genitourinary Cancer Patients That Suffered COVID-19
Started | 410
Completed | 410
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Genitourinary Cancer Patients That Suffered COVID-19
Number analyzed (Participants) | 408
Age, Continuous [Median (Full Range); unit: years] | 70 [17 to 100]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 357
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 408
  More than one race | 0
  Unknown or Not Reported | 0
Smoking status [Count of Participants; unit: Participants]
  Never | 136
  Ever | 231
  UK | 41
Comorbities [Count of Participants; unit: Participants]
  Hypertension | 224
  Diabetes | 92
  Cardiopathy | 79
  COPD / Asma | 57
  Hepatopathy | 19
  Nephropathy | 53
  None | 121
Cancer type [Count of Participants; unit: Participants]
  Prostate | 166
  Urothelial | 128
  Kidney | 90
  Testicular | 23
  Penile | 1
Clinical cancer stage at cancer diagnosis; [Count of Participants; unit: Participants] — Cancer staging measures the extent of spread of the disease. This scale is established by the American Joint Committee in Cancer (AJCC). The categories range from localized / regional tumours (Stage I-II) to locally advanced (Stage III) or metastatic (Stage IV)
  Participants
    0 | 2
    I | 54
    II | 64
    III | 90
    IV | 166
    UK | 32
Time from cancer diagnosis to SARS-CoV-2 infection [Median (Full Range); unit: months] | 32 [27 to 38]
Clinical cancer stage at SARS-CoV-2 infection [Count of Participants; unit: Participants] — Cancer staging measures the extent of spread of the disease. This scale is established by the American Joint Committee in Cancer (AJCC). The categories range from localized / regional tumours (Stage I-II) to locally advanced (Stage III) or metastatic (Stage IV)
  Participants
    o | 24
    I | 19
    II | 22
    III | 29
    IV | 291
    UK | 23
Histopathological grade at SARS-CoV-2 infection [Count of Participants; unit: Participants]
  Well differentiated | 31
  Moderately differentiated | 61
  Poorly differentiated | 136
  UK | 180
Anticancer treatment status at SARS-CoV-2 infection [Count of Participants; unit: Participants]
  Active | 238
  Follow-up | 170
Anticancer treatment type at SARS-CoV-2 infection [Count of Participants; unit: Participants]
  Neo-adjuvant | 8
  Adjuvant | 10
  Metastatic / palliative | 219
  UK | 1

OUTCOME MEASURES:

1. Primary Outcome: Age at Baseline
Description: Describe the population infected by COVID-19 with genitourinary tumors (urothelial cancer, prostate cancer, testicular cancer and kidney cancer) treated in Spanish hospitals, know the clinical presentation: Spcifically here we reported the Age
Time Frame: Baseline, at the time of inclusion
Population: Describe the population infected by COVID-19 with genitourinary tumors (urothelial cancer, prostate cancer, testicular cancer and kidney cancer) treated in Spanish hospitals
Measure: Median (Full Range); unit: years
Arm/Group | Genitourinary Cancer Patients That Suffered COVID-19
Number analyzed (Participants) | 408
years | 70 [17 to 100]

2. Primary Outcome: Frequency of Complications of COVID-19 Intercurrent Infection
Description: Percentage of patients with complications associated to COVID-19 infection (classified by type and severity)
Time Frame: Through study completion, average 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Genitourinary Cancer Patients That Suffered COVID-19
Number analyzed (Participants) | 408
Participants
  Death secondary to infectioninfection | 73
  ICU admission due to need of symptom control | 5
  Hospital admission due to need of symptom control | 136
  Need for mechanical ventilation | 3
  No complications. Common infection at home | 191

3. Primary Outcome: Frequency of Complications of COVID-19 Infection (Pneumonia) Stratified by Treatment
Description: To assess the possible relationship of the different oncological treatments administered to these patients with the clinical evolution of the COVID-19 infection. Complications will be classified by type and severity in groups of patients stratified by the oncological treatment received.
Time Frame: Through study completion, average 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Genitourinary Cancer Patients That Suffered COVID-19
Number analyzed (Participants) | 408
Participants
  Immunotherapy treatment/no Pneumonia | 51
  Immunotherapy treatment/ Pneumonia | 36
  No Immunotherapy treatment/no Pneumonia | 181
  No Immunotherapy treatment/Pneumonia | 140

4. Primary Outcome: Frequency of Complications of COVID-19 Infection in Patients With Genitourinary Cancer Stratified by Anti-androgenic Oncological Treatment
Description: To evaluate in patients with Genitourinary Cancer the impact of androgen deprivation therapy (ADT) and new antiandrogenic agents (NAH) with or without corticosteroids on the infection COVID-19 as mean of frequency in complications of COVID-19 infection classified by type and severity
Time Frame: Through study completion, average 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Genitourinary Cancer Patients That Suffered COVID-19
Number analyzed (Participants) | 408
Participants
  Corticosteroid treatment/ no Pneumonia | 59
  Corticosteroid treatment/ si Pneumonia | 55
  No Corticosteroid treatment/ no Pneumonia | 173
  No Corticosteroid treatment/ si Pneumonia | 120
  UK | 1

5. Primary Outcome: Frequency of Complications of COVID-19 Infection Stratified by Treatment (Immunotherapy vs no Immunotherapy)
Description: as for outcome 3
Time Frame: Through study completion, average 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Genitourinary Cancer Patients That Suffered COVID-19
Number analyzed (Participants) | 408
Participants
  Immunotherapy treatment /no complications | 45
  Immunotherapy treatment /admissions | 31
  Immunotherapy treatment /Death secondary to infection | 11
  No Immunotherapy treatment /no complications | 146
  No Immunotherapy treatment /admissions | 113
  No Immunotherapy treatment /Death secondary to infection | 62

6. Primary Outcome: Frequency of Adverse Events Related to Immunotherapy Targeted to Cancer (Classified by Type and Severity)
Description: To specifically assess the impact of COVID-19 infection on the toxicity of immunotherapy treatment (mainly pneumonitis) and the impact of immunotherapy on the evolution of the infectious picture in patients with tumors of genitourinary origin. three different scenarios: during treatment, after treatment and in patients who receive treatment after the infection has passed.
Time Frame: Through study completion, average 1 year. Measured at 3 scenarios (during treatment, after treatment and therapies indicated after infection has passed)
Measure: Count of Participants; unit: Participants
Groups:
- Patients Diagnosed With Genitourinary Cancer Hat Suffered COVID-19 Treatment With Immunotherapy: Patients diagnosed with genitourinary cancer (urothelial, kidney, prostate and germ) that suffered from COVID-19 infection prior to cancer treatment, during treatment, or after treatment with immunotherapy
Arm/Group | Patients Diagnosed With Genitourinary Cancer Hat Suffered COVID-19 Treatment With Immunotherapy
Number analyzed (Participants) | 87
Participants
  Arthritis G1 | 1
  Arthritis G3 | 1
  Colitis G1 | 1
  Colitis G2 | 1
  Colitis G3 | 1
  Hepatitis G2 | 3
  Hepatitis G3 | 3
  Hepatitis G4 | 1
  Hypophysitis G2 | 1
  Nephritis G1 | 1
  Nephritis G2 | 1
  Nephritis G3 | 1
  Nephritis G4 | 1
  Pneumonitis G2 | 1
  Thyroiditis G1 | 2
  Thyroiditis G2 | 2

7. Secondary Outcome: COVID-19 Mortality Rate in Patients With Genitourinary Cancer
Description: To assess the mortality associated with COVID-19 infection in the population with genitourinary tumors. Percentage of patients alive / dead at discharge.
Time Frame: Through study completion, average 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Genitourinary Cancer Patients That Suffered COVID-19
Number analyzed (Participants) | 408
Participants
  Alive | 137
  Dead | 80
  NA | 191

8. Secondary Outcome: COVID-19 Complication Rate in Patients With Genitourinary Cancer
Description: Evaluate the rate (percentage) of complications that have required hospital admission and / or ICU treatment. Complications will be classified by type and severity and represented as percentage of patients presenting them.
Time Frame: Through study completion, average 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Genitourinary Cancer Patients That Suffered COVID-19
Number analyzed (Participants) | 408
Participants
  Death secondary to infection | 73
  ICU admission due to need of symptom control | 5
  Hospital admission due to need of symptom control | 136
  Need for mechanical ventilation | 3
  No complications. Common infection at home | 191

9. Secondary Outcome: Asymptomatic Rate
Description: Describe the frequency of asymptomatic or minimally symptomatic COVID-19 infections.
Time Frame: Through study completion, average 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Genitourinary Cancer Patients That Suffered COVID-19
Number analyzed (Participants) | 408
Participants
  symptomatic | 308
  Asymptomatic | 100

10. Secondary Outcome: Asymptomatic Rate in Renal Cancer
Description: Describe the frequency of asymptomatic or minimally symptomatic COVID-19 infections.
Time Frame: Through study completion, average 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Renal Cancer Patients That Suffered COVID-19: Patients diagnosed with renal cancer that suffered from COVID-19 infection prior to cancer treatment, during treatment, or after treatment.
Arm/Group | Renal Cancer Patients That Suffered COVID-19
Number analyzed (Participants) | 90
Participants
  Symptomatic | 63
  Asymptomatic | 27

11. Secondary Outcome: Asymptomatic Rate in Urothelial Cancer
Description: Describe the frequency of asymptomatic or minimally symptomatic COVID-19 infections.
Time Frame: Through study completion, average 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Urothelial Cancer Patients That Suffered COVID-19: Patients diagnosed with urothelial cancer that suffered from COVID-19 infection prior to cancer treatment, during treatment, or after treatment.
Arm/Group | Urothelial Cancer Patients That Suffered COVID-19
Number analyzed (Participants) | 128
Participants
  Asymptomatic | 32
  Symptomatic | 96

12. Secondary Outcome: Asymptomatic Rate in Prostate Cancer
Description: Describe the frequency of asymptomatic or minimally symptomatic COVID-19 infections
Time Frame: Through study completion, average 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Prostate Cancer Patients That Suffered COVID-19: Patients diagnosed with prostate cancer that suffered from COVID-19 infection prior to cancer treatment, during treatment, or after treatment.
Arm/Group | Prostate Cancer Patients That Suffered COVID-19
Number analyzed (Participants) | 166
Participants
  Asymptomatic | 33
  Symptomatic | 133

13. Secondary Outcome: Asymptomatic Rate in Testicular Cancer
Description: Describe the frequency of asymptomatic or minimally symptomatic COVID-19 infections
Time Frame: Through study completion, average 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Testicular Cancer Patients That Suffered COVID-19: Patients diagnosed with testicular cancer that suffered from COVID-19 infection prior to cancer treatment, during treatment, or after treatment.
Arm/Group | Testicular Cancer Patients That Suffered COVID-19
Number analyzed (Participants) | 21
Participants
  asymptomatic | 6
  symptomatic | 15

14. Secondary Outcome: Frequency of Delays/Modifications on Cancer Treatment Schedule
Description: delays / modifications in cancer follow-up or treatment regimens.
Time Frame: Through study completion, average 1 year
Population: Patients with genitourinary tumor presenting Covid-19 infection with prospective part who start/restart treatment
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Genitourinary Tumor Presenting Covid-19 Infection With Prospective Part: Patients with prospective part
Arm/Group | Patients With Genitourinary Tumor Presenting Covid-19 Infection With Prospective Part
Number analyzed (Participants) | 326
Participants
  Start Treatment after COVID-19 | 20
  Restart Treatment after COVID-19 | 146
  With treatment after COVID-19 without specifying start/restart | 6
  Without oncology treatment after COVID-19 (reported) | 154

15. Secondary Outcome: Frequency of Delays/Modifications on Cancer Treatment Schedule
Description: delays / modifications in cancer follow-up or treatment regimens.
Time Frame: Through study completion, average 1 year
Population: Patients with genitourinary tumor presenting Covid-19 infection with prospective part witn treatment modifications
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Genitourinary Tumor Presenting Covid-19 Infection With Prospective Part: Patients with genitourinary tumor presenting Covid-19 infection with treatment modifications in cancer follow-up or treatment regimens.
Arm/Group | Patients With Genitourinary Tumor Presenting Covid-19 Infection With Prospective Part
Number analyzed (Participants) | 38
Participants
  Dose | 1
  Change in administration schedule | 15
  Temporary suspension of treatment | 22

16. Secondary Outcome: Frequency of Delays/Modifications on Cancer Treatment Schedule
Description: delays / modifications in cancer follow-up or treatment regimens.
Time Frame: Through study completion, average 1 year
Population: Patients with genitourinary tumor presenting Covid-19 infection with prospective part
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Genitourinary Tumor Presenting Covid-19 Infection With Prospective Part
Number analyzed (Participants) | 326
Participants
  Yes Treatment modification (prospective visit) | 38
  No Treatment modification (prospective visit) | 108
  New treatment o no treatment start date | 24
  NA/UK | 156

17. Secondary Outcome: Progression Free Survival in Patients With Genitourinary Tumors That Suffered COVID-19, Patients With a First Line Treatment Ongoing at the Moment of COVID Infection
Description: It is expected to obtain data on time to progression and overall survival of cancer patients, which can be compared with the reference values for each type of tumor pathology.
  PROGRESSION FREE SURVIVAL (FIRST LINE IN METASTATIC OR ADVANCED SETTING) The date of treatment start (treatment ongoing at the moment of COVID infection) is taken as the start date of follow-up. Only patients with a first line treatment ongoing at the moment of COVID infection were analyzed.
Time Frame: From start of treatment until progression or death, up to 130 months
Population: Patients with genitourinary tumors that suffered COVID-19. Only patients with a first line treatment ongoing at the moment of COVID infection were analyzed.
Measure: Mean (95% Confidence Interval); unit: months
Groups:
- Genitourinary Cancer Patients With a First Line Treatment Ongoing at the Moment of COVID Infection.: Patients diagnosed with genitourinary cancer (urothelial, kidney, prostate and germ) that suffered from COVID-19 infection with a first line treatment ongoing at the moment of COVID infection were analyzed.
Arm/Group | Genitourinary Cancer Patients With a First Line Treatment Ongoing at the Moment of COVID Infection.
Number analyzed (Participants) | 56
months
  Renal: number analyzed (Participants) | 23
  Renal | 93.26 [45.62 to 140.91]
  Urothelial: number analyzed (Participants) | 14
  Urothelial | 80.13 [28.38 to 131.88]
  Prostate: number analyzed (Participants) | 19
  Prostate | 121.94 [96.68 to 147.2]

18. Secondary Outcome: Overall Survival in Patients With Genitourinary Tumors That Suffered COVID-19
Description: It is expected to obtain data on time to progression and overall survival of cancer patients, which can be compared with the reference values for each type of tumor pathology.
  For the calculation of overall survival, it is taken from the date of cancer diagnosis to the date of death (at any time, not only in a prospective part).
Time Frame: From start of treatment until progression or death, up to 130 months
Population: Patients with genitourinary tumor presenting Covid-19 infection with prospective part
Measure: Mean (95% Confidence Interval); unit: years
Arm/Group | Patients With Genitourinary Tumor Presenting Covid-19 Infection With Prospective Part
Number analyzed (Participants) | 405
years
  Renal: number analyzed (Participants) | 90
  Renal | 18.36 [14.51 to 22.22]
  Urothelial: number analyzed (Participants) | 128
  Urothelial | 7.03 [4.91 to 9.14]
  Prostate: number analyzed (Participants) | 166
  Prostate | 11.49 [9.85 to 13.13]
  Testicular: number analyzed (Participants) | 21
  Testicular | 24.37 [19.97 to 28.76]

ADVERSE EVENTS:
Time Frame: 2 year Note: Adverse events were only collected and reported by those patients on active immunotherapy by the time of SARS-CoV-2 infection (n=87)
Description: Adverse events were only collected and reported in the subgroup of patients treated with immunotherapy (n=87) All cause mortality reported in the overall population
Groups:
- Adverse Events: Adverse events reported by those patients on active immunotherapy by the time of SARS-CoV-2 infection.
  The main scope of this trial was not safety. Therefore, the study did not record adverse events in patients treated with other therapies. The study did not record serious adverse events sistematically.
  This partial information about safety was the only information of adverse events collected during this observational study.
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 152/408
Serious Adverse Events (participants affected / at risk) | 0/87
Other Adverse Events (participants affected / at risk) | 22/87
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adverse Events (N=87)
Hepatitis (Hepatobiliary disorders) | 7
Nephritis (General disorders) | 4
Thyroiditis (Endocrine disorders) | 4
Colitis (Infections and infestations) | 3
Arthritis (General disorders) | 2
Pneumonitis (Infections and infestations) | 1
Hypophysitis (Endocrine disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT04578132/Prot_SAP_000.pdf